CLINICAL TRIAL: NCT03861741
Title: A Study to Evaluate the Feasibility of Screening Relatives of Patients Affected by Non-Syndromic Thoracic Aortic Diseases: The ReST Study
Brief Title: A Study to Evaluate the Feasibility of Screening Relatives of Patients Affected by Non-Syndromic Thoracic Aortic Diseases
Acronym: ReST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0676
Record Dates: First submitted 2019-02-18; First posted 2019-03-04 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Screening; Aortic Aneurysm and Dissection; Genetic Disease
Keywords: screening, aortic disease, mortality, genetic testing, imaging
MeSH Terms: conditions — Aortic Dissection; Genetic Diseases, Inborn; Aortic Diseases | interventions — Exome Sequencing; Magnetic Resonance Imaging; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: This pilot study will recruit relatives of 16 patients with a diagnosis of non-syndromic thoracic aortic disease. As many FDR and SDR of the proband (index patient) as possible will be recruited into the study (family based analysis). They will be screened through complete clinical evaluations, genetic tests (whole exome sequencing) and imaging modalities (TTE and MRI) for the presence of newly NS-TADs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): All participants will be screened through complete clinical evaluations, genetic tests and imaging modalities (TTE and MRI) for the presence of newly Non Syndromic-Thoracic Aortic Diseases. Demographic and clinical data from all participants will be collected using case report forms, and by accessing their medical records. Data on imaging investigations will be obtained from TTE and MRI. Blood samples will be used for the purpose of isolation of genetic material and subsequent whole exome sequencing along with the analysis of selected loci. Additional citrated blood samples and plasma will be collected and stored for the potential analysis of circulating microvesicles and miRNA.
  Interventions: Genetic: WES; Diagnostic Test: MRI; Diagnostic Test: TTE; Other: Questionnaire

INTERVENTIONS:
Genetic: WES — A peripheral venous blood sample will be processed internally, and externally subjected to WES. Only genetic material from relatives of probands in which a mutation has been identified will be sequenced.
  Other Names: Whole exome sequencing
Diagnostic Test: MRI — A MRI of the thoracic aorta will be performed in all relatives able to attend the Glenfield Hospital and who have no contra-indications to this imaging modality; pulse-wave velocity will be recorded.
  Other Names: Magnetic resonance imaging
Diagnostic Test: TTE — TTE screening will be performed by a trained physiologist. Aortic diameter will be measured from the parasternal long-axis view at the sinuses of Valsalva and at the widest level of the ascending aorta. All measurements will be made in end-diastole.
  Other Names: Trans-thoracic echocardiography
Other: Questionnaire — Acceptability questionnaires will be submitted to assess a baseline score of depression/anxiety that will be compared with a follow up value at three months

SUMMARY:
The primary hypothesis is that a tailored programme of genetic and imaging screening of first- and second-degree relatives of patients affected by non-syndromic forms of thoracic aortic diseases will identify individuals at risk of death from these conditions. These individuals would constitute specific population of patients, requiring dedicated imaging surveillance and/or earlier prophylactic aortic surgery.

DETAILED DESCRIPTION:
Diseases involving the thoracic aorta (the major artery in the body) are a major health problem affecting an increasing number of people worldwide.

In particular, a group of these conditions termed Non-Syndromic Aortic Diseases (NS-TAD), can develop without any obvious symptoms or external features which prevents early identification. Unfortunately, if not treated, the aorta may enlarge and lead to dissection, a life-threatening medical emergency. For this reason, the investigators believe it might be helpful to investigate relatives of patients undergoing surgery for thoracic aortic disease to understand if there are tests that could help identify and treat this condition at the right time.

Therefore the investigators propose to conduct a feasibility study to identify the practical issues and challenges that would need to be overcome in order to perform a successful tailored genetic (by collecting a small blood sample) and imaging (with exams such as echocardiography and MRI) screening in such population of individuals.

Moreover, all participants will receive two questionnaires to ask their opinion about the study and to measure their levels of anxiety and depression, to judge whether and how this study has affected their emotional status.

The study will be carried out at the Department of Cardiovascular Sciences Glenfield Hospital, University Hospitals of Leicester NHS Trust.

ELIGIBILITY:
Inclusion Criteria:

1. NS-TAD probands operated on (n=16).
2. FDR and SDR, aged 16 and above:

   1. At least two relatives willing to participate in the screening programme.
   2. Relatives able to understand English.

Exclusion Criteria:

1. Probands with syndromic aortopathies, including Marfan Syndrome, Loeys-Dietz Syndrome, Ehlers-Danlos Syndrome, Shprintzen-Goldberg syndrome, aneurysm-osteoarthritis syndrome, arterial tortuosity syndrome, and cutis laxa syndrome.
2. Probands with aortic lesions associated with trauma and infections.
3. Probands/relatives unable to give informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-05-20 (Estimated)

PRIMARY OUTCOMES:
Rate of genetic diagnosis | Through study completion, an average of 1 year
  Frequency of first and second degree relatives with newly identified genetic loci associated with NS-TADs.
Rate of diagnosis through imaging modalities | At the end of recruitment stage, an average of 6 months
  Frequency of newly diagnosed TAD through imaging modalities in first- and second-degree relatives of probands affected by NS-TADs.

SECONDARY OUTCOMES:
Genetic variants | Through study completion, an average of 1 year
  Genetic variants associated with NS-TADs, identified from a panel of 55 loci, and rate of identification of each mutation.
Family rate of genetic carriers | Through study completion, an average of 1 year
  Rate of genetic carriers in each affected family.
Penetrance | Through study completion, an average of 1 year
  Genetic penetrance of the NS-TADs (proportion of individuals carrying a particular variant of a gene that are also affected by NS-TAD).
Mode of inheritance | Through study completion, an average of 1 year
  Pattern of inheritance of the NS-TADs.
Male: female preponderance | Through study completion, an average of 1 year
  Male: female preponderance of NS-TADs.
Aortic Compliance | Imaging tests completion, an average of 6 months.
  Measured as an MRI feature of affected and unaffected thoracic aortas.
Aortic Distensibility | Imaging tests completion, an average of 6 months.
  Measured as an MRI feature of affected and unaffected thoracic aortas.
Rates of concomitant external and cardiovascular characteristics | Baseline clinical assessment
  Rates of concomitant cardiovascular diseases (e.g. patent ductus arteriosus, cerebrovascular aneurysm) and external physical features (e.g. pectus excavates, livedo reticularis).
Response rate | Baseline clinical assessment
  Response rates (recruitment) among the probands and their relatives.
Acceptability questionnaires | Baseline and 3 months follow up
  Semi-quantitative evaluation of the participant experience awareness and acceptability of the screening and consent process, obtained by questionnaires administered to the patients and relatives.
  Scales will be composed by 10 items, each can be rated with a score from 1 to 5. No threshold will be preset. Descriptive statistics will be used to present the results.
Depression evaluation | Baseline and 3 months follow up
  Semi-quantitative evaluation of the impact of the screening process on depression in probands and their relatives (baseline and 3 months), based on Patient Health Questionnaire (PHQ-9) score. Score range goes from 0 to 27, proposed cut-off for active treatment is 15.
Anxiety evaluation | Baseline and 3 months follow up
  Semi-quantitative evaluation of the impact of the screening process on anxiety in probands and their relatives (baseline and 3 months), based on Generalized Anxiety Disorder (GAD-7) score. Score range goes from 0 to 21, proposed cut-off for further assessment is 10.
Health-related Quality of Life evaluation | Baseline and 3 months follow up
  Semi-quantitative evaluation of the impact of the screening process on health-related quality of life in probands and their relatives (baseline and 3 months), based on Short Form (36) Health Survey (SF-36) score. Said questionnaire is made up of eight scales, which are the weighted sums of the items for each section; a score of zero corresponds to maximum disability while 100 correlates to no disability.
Resource use of genetic screening | 3 months follow up
  Resource uses in terms of unitary costs of the genetic screening process.
Resource use of imaging screening | 3 months follow up
  Resource uses in terms of unitary costs of the imaging screening process.
Resource use (hospital visits) | 3 months follow up
  Number of participants reaching the research centre.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin J Murphy, Prof, Principal Investigator — University of Leicester; Giovanni Mariscalco, Prof, Principal Investigator — University of Leicester
Locations (1):
- Department of Cardiovascular Sciences, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mariscalco G, Debiec R, Elefteriades JA, Samani NJ, Murphy GJ. Systematic Review of Studies That Have Evaluated Screening Tests in Relatives of Patients Affected by Nonsyndromic Thoracic Aortic Disease. J Am Heart Assoc. 2018 Aug 7;7(15):e009302. doi: 10.1161/JAHA.118.009302. PMID 30371227
- [Derived] Abbasciano RG, Mariscalco G, Barwell J, Owens G, Zakkar M, Joel-David L, Pathak S, Adebayo A, Shannon N, Haines RL, Aujla H, Eagle-Hemming B, Kumar T, Lai F, Wozniak M, Murphy G. Evaluating the Feasibility of Screening Relatives of Patients Affected by Nonsyndromic Thoracic Aortic Diseases: The REST Study. J Am Heart Assoc. 2022 Apr 19;11(8):e023741. doi: 10.1161/JAHA.121.023741. Epub 2022 Apr 6. PMID 35383466

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/41/NCT03861741/SAP_000.pdf